CLINICAL TRIAL: NCT06031870
Title: Beckenboden-Rehabilitationsstudie (BREST)
Brief Title: Pelvic Floor Rehabilitation Study (Beckenboden-Rehabilitationsstudie - BREST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Soren Lange, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-13832
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Postpartum Urinary Incontinence
MeSH Terms: interventions — Pessaries; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (Active Comparator)
  Interventions: Behavioral: Standard care
- Pelvic floor muscle training (Active Comparator)
  Interventions: Procedure: Pelvic floor muscle training
- Vaginal pessary (Experimental)
  Interventions: Device: Vaginal pessary

INTERVENTIONS:
Device: Vaginal pessary — In the pessary group, all patients received a cube pessary, which was individually adapted to each patient. These pessaries exist in sizes 0 (25 mm edge length) to 9 (75 mm edge length). Patients were instructed by a physician or a trained nurse on how to autonomously manage the pessary, including daily changing and cleaning. After one week of treatment, all patients had an office visit to check if fitting was correct and if autonomous handling of the pessary was feasible. Treatment duration was 12 weeks.
  Arms: Vaginal pessary
Behavioral: Standard care — Standard care consisted of a pelvic floor group exercise course led by a midwife, a physiotherapist, or an osteopath. Courses were in general once a week for a minimum of seven to a maximum of twelve weeks. The course was chosen by the patient, and the study team had no influence on the choice.
  Arms: Standard care
Procedure: Pelvic floor muscle training — Twelve pelvic floor physiotherapy sessions were prescribed by the study physician. Pelvic floor physiotherapy was performed in individual courses by trained physiotherapists. The patient was free to choose the physiotherapist and the study team had no influence on the choice.
  Arms: Pelvic floor muscle training

SUMMARY:
This study compares the effectiveness of standard care, pelvic floor muscle training or vaginal pessary for the treatment of postpartum urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* gave birth within the 12 weeks prior to the postpartum visit
* postpartum urinary incontinence
* able to understand and give consent in German

Exclusion Criteria:

* treatment for postpartum urinary incontinence that started prior to inclusion
* any neurologic disease that impairs bladder function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
patients' self-reported satisfaction with the treatment | 12 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Die GynPraxis, Alzey
  - Die GynPraxis, Bad Kreuznach
  - Die GynPraxis, Lampertheim
  - Die GynPraxis, Mainz

IPD SHARING:
Plan to Share IPD: Undecided